CLINICAL TRIAL: NCT04346446
Title: Efficacy of Convalescent Plasma Therapy in Severely Sick COVID-19 Patients: A Pilot Randomized Controlled Trial
Brief Title: Efficacy of Convalescent Plasma Therapy in Severely Sick COVID-19 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-COVID-02
Record Dates: First submitted 2020-04-14; First posted 2020-04-15 (Actual); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: COVID
Keywords: convalescent plasma,COVID,SARS-COV -2
MeSH Terms: interventions — Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent Plasma+Supportive Care (Experimental): Convalescent Plasma+Supportive Care Convalescent plasma from recovered COVID-19 patients will be transfused to severely sick COVID-19 infected patients
  Interventions: Drug: Convalescent Plasma Transfusion; Other: Supportive Care
- Random Donor Plasma+Supportive Care (Active Comparator): Random Donor Plasma+Supportive Care
  Interventions: Other: Supportive Care; Drug: Random Donor Plasma

INTERVENTIONS:
Drug: Convalescent Plasma Transfusion — Convalescent Plasma Transfusion
  Arms: Convalescent Plasma+Supportive Care
Other: Supportive Care — Supportive Care
Drug: Random Donor Plasma — Random Donor Plasma will be transfuse from 200 to 600 mL according to the patient requirement
  Arms: Random Donor Plasma+Supportive Care

SUMMARY:
Currently, no effective treatments are available for the COVID-19 pandemic, which is related to more than 70,000 deaths all over the world. Scientists and Researchers are working on many aspects of treatment options for the development of vaccination and medication to combat this life-threatening problem. Convalescent plasma from recovered COVID-19 patients contains antibodies against COVID-19 which may be beneficial to severely sick COVID019 infected patients. We have planned a randomized controlled trial to assess the efficacy of this therapy in COVID-19 infected sick patients. We will collect up to 500 ml Convalescent Plasma from the COVID-19 infected recovered patient after 14 days of clinical and radiological recovery with two consecutive COVID-19 negative tests by PCR. We will further test the sample from the collected plasma for COVID-19 specific antibodies and their titer. This plasma will be frozen and sent to the treating center (MAMC). 200-600 ml of convalescent plasma will be transfused to patients who fit the eligibility criteria and are randomized to the convalescent plasma group. This will be done in severely sick patients. Data will be collected for the benefit and adverse events related to convalescent plasma transfusion.

DETAILED DESCRIPTION:
For Donors:

Microtiter plates will be coated overnight at 4°C with 4 μg/mL recombinant SARS-CoV-2 RBD (receptor binding domain) proteins (50 μL per well). The plates will be washed 3 times with phosphate-buffered saline (PBS) containing 0.1% vol/vol Tween-20(PBST) and blocked with blocking solution (PBS containing 2% wt/vol nonfat dry milk) for 2 hours at 37 °C. The plates will be then washed with PBST. The serum samples will be diluted to 200-fold into PBS as initial concentration, and serial 3-fold dilutions of serum will be added to the wells and incubated at 37 °C for 60 minutes. After 3 washes, 100 μL of horseradish peroxidase-conjugated goat anti-human IgG (for IgG antibody titer detection)and IgM (for IgM antibody titer detection) antibodies solution will be added to each plate, respectively, and incubated at 37 °C for 60 minutes. After 5 washes, 100 μL of tetramethylbenzidine substrate will be added at room temperature in the dark. After 15 minutes, the reaction will be stopped with a2MH2SO4 solution (sulfuric acid). The absorbance will be measured at 450nm. All samples will be run in triplicate. The IgG titers will be determined by endpoint dilution.

Serum Neutralization Assay Vero cells (104) will be seeded 24 hours before the infection in a 96-well plate. On the day of infection, the cells will be washed twice. Serum samples from patients will be incubated at 56 °C for 30 minutes and then diluted 2-fold in cell culture medium (modified eagle medium). Aliquots (40 μL) of diluted serum samples (from2-fold to 2056-fold) will be added to 50 μL of cell culture medium containing 50 times the tissue culture infective dose (TCID50) of the virus strain on a 96-well plate and incubated at 37 °C for 2 hours in CO2 5% vol/vol. Virus antibody mix will be added to cells in 96-well plates and plates will be incubated at 37 °C with a microscopic examination for cytopathic effect after 5-day incubation. The highest dilution of serum that showed inhibition activity of SARS-CoV-2 will be recorded as the neutralizing antibody titer. Assays will be performed in triplicate with negative control samples from healthy volunteers.

For recipients:

The serum of each recipient will be obtained and enzyme-linked immunosorbent assay (ELISA) and neutralizing antibody titers will be tested one day prior to the convalescent plasma transfusion. Changes of Receptor Binding Domain-Specific IgG titre and neutralizing antibody titers before and after convalescent plasma transfusion in patients will be obtained on day 0, day 1, day 3 and day 7. if possible.

All included patients would be randomized to receive either standard medical therapy (supportive therapy) with random donor plasma versus convalescent plasma and standard medical therapy Clinical information of all enrolled patients including symptoms at presentation, time to presentation to the hospital and development of pulmonary symptoms would be recorded. The details of comorbid diseases as measured by the Charlson index of comorbidity and Acute Physiology and Chronic Health Evaluation II (APACHE II). Details of cross-sectional imaging, chest-x-ray, bacterial or fungal co-infections and details of antibiotic treatment would be recorded. Development of complications including acute kidney injury, acute coronary syndrome, myocarditis, acute respiratory distress syndrome, and nosocomial infection will be recorded. The use of high-flow oxygen, non-invasive and invasive ventilation will follow standard guidelines and will be recorded. The details of antiviral treatment including oral oseltamivir, hydroxychloroquine, and use of intravenous steroids will be recorded for all enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

-

Recipient:

Severe COVID -19 infections defined as WHO Interim Guidance and the Guideline of Diagnosis and Treatment of COVID-19 of National Health Commission of China (version 5.0) with confirmation by real-time RT-PCR assay with severe disease i.e. meeting any 2 of the following criteria-

1. Respiratory distress, RR ≥30 beats/min
2. Oxygen saturation level less than 93% in resting state
3. Partial pressure of oxygen (PaO2)/oxygen concentration (FiO2) ≤ 300 mmHg.
4. Lung infiltrates > 50% within 24 to 48 hours
5. Very sick (on ventilator) and patients with co-morbidities such as patients with known co-morbid diseases (COPD, CAD, CLD, CKD, cardiopulmonary disease-structural or valvular heart disease)
6. Patient presenting with multi organ failure or requiring mechanical ventilation.

Donor:

* Known case of recovered COVID-19 Infection, and
* Complete resolution of symptoms at least 28 days prior to donation or Complete resolution of symptoms at least 14 days prior to donation and negative results for COVID-19 either from one or more nasopharyngeal swab specimens or by a molecular diagnostic test from the blood, And Negative RT-PCR for COVID-19 on two sequential paired nasopharyngeal and throat specimens > 24 hrs apart (WHO-CDC guideline).
* Donor Plasma after 2 negative tests and 2 weeks of remaining asymptomatic, without antibody titre & presence of IgG/IgM antibodies to COVID-19 by serological as per manufacturers instructions. Donors negative for these will be deferred).
* Fulfill all criteria of donor eligibility for donor Plasmapheresis under the Drugs & Cosmetics Act and Rules 1945, amended 11.03.2020.

Exclusion Criteria:

- Recipient

* Patients with age less than 18 years.
* Pregnancy
* Individual with HIV and Hepatitis
* Morbid Obesity BMI>35 kg/m2
* Extremely moribund patients with an expected life expectancy of less than 24 hours.
* Failure to give informed consent from the patient or family members.
* Hemodynamic instability requiring vasopressors.
* Previous allergic history to plasma.

Donor:

* Donors age < 18 & ≥60 years old
* Do not fulfil all criteria of donor eligibility for donor Plasmapheresis under the Drugs & Cosmetics Act and Rules 1945, amended 11.03.2020.
* Females who have been pregnant and previously transfused donors (to prevent TRALI).
* Donors who have taken steroids during treatment for COVID-19.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Proportion of patients remaining free of mechanical ventilation in both groups | Day 7

SECONDARY OUTCOMES:
Mortality in both groups | Day 28
Improvement in Pa02/Fi02 ratio in both groups | Day 2
Improvement in Pa02/Fi02 ratio in both groups | Day 7
Improvement in SOFA score in both groups | Day 2
Improvement in SOFA score in both groups | Day 7
Duration of hospital Stay in both group. | Day 28
Duration of Intensive Care Unit stay in both groups. | Day 28
Requirements of Vasopressor in both groups. | Day 28
Days free of dialysis in both groups. | Day 28

CONTACTS AND LOCATIONS:
Locations (2):
- India (2):
  - Maulana Azad medical College, New Delhi, National Capital Territory of Delhi
  - Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969